CLINICAL TRIAL: NCT04427176
Title: Evaluation of ARFC Masks Equipped With CF5 Filter in the Care Unit to Allow a Wider Distribution of FFP2 Masks (Covid-19).
Acronym: Masq-Aute
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 20CH073; 2020-A00817-32 (Other: ANSM)
Record Dates: First submitted 2020-06-10; First posted 2020-06-11 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Nurse
Keywords: mask; ARFC; Covid-19; protection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nurses: Nursing staff working 8 or 12 hours a day for 2 consecutive days in a COVID unit at the hospital of Saint Etienne will be included.
  They will be wear ARFC mask.
  Interventions: Device: ARFC mask

INTERVENTIONS:
Device: ARFC mask — Nurse will wear the ARFC mask during working days. The total duration of the study will be 48 hours for each participant, 2 consecutive working days of 8 or 12 hours.

SUMMARY:
The current outbreak of Covid-19 requires the wearing of FFP2 respiratory protective devices by healthcare personnel to limit their contamination.

However, there is currently a shortage of masks in France due to insufficient national stocks while the disease is spreading.

There is an urgent need to save FFP2 masks to enable healthcare personnel to continue to provide care in complete safety. Contamination of staff due to insufficient masks would have consequences by limiting access to care for infected patients and putting caregivers at potential risk of death. Caregiver protection is also intended to contain the risk of nosocomial epidemics. We propose the use of ARFC masks by Covid-19+ units. These ARFC masks provide optimal security against the risk of aerosolization of contaminated biological liquids. They are masks modified to be usable by civilians, resulting from the technology of combat masks, specially designed for use in NRBC (Nuclear, Radiological, Biological and Chemical) atmosphere.

ELIGIBILITY:
Inclusion Criteria:

* Nursing staff working 8 or 12 hours a day for 2 consecutive days in a COVID unit at the hospital of Saint Etienne.
* Subjects affiliated to or entitled to a social security scheme
* Subject who received informed information about the study and agreed to participate in the study

Exclusion Criteria:

* Allergy to ARCF mask material: polyurethane
* Impossibility of supporting a tight mask on the face
* Potential contraindication to wearing a mask, such as the existence of claustrophobia
* Beard and moustache wearer
* Suspicion of COVID-19 infection
* Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nursing staff working 8 or 12 hours a day for 2 consecutive days in a COVID unit at the hospital of Saint Etienne.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Evaluate the feasibility of the use of an ARFC mask by nursing staff, in terms of tolerance | Hour: 48
  Tolerance will be assessed by the nursing staff by means of a visual analogue scale from 0: no tolerance to 10: perfect tolerance. It will be evaluated 48 hours after the inclusion.
Evaluate the feasibility of the use of an ARFC mask by nursing staff, in terms of compatibility with technical gestures. | Hour: 48
  Compatibility will be assessed by the number of catheter insertion and blood sampling failures in relation to the total number of catheter insertions and blood sampling indicated at 48 hours after the inclusion.

SECONDARY OUTCOMES:
Assess the acceptability of the wearing of an ARFC mask by nursing staff | Hours: 0, 48
  To compare acceptability questionnaires complete at inclusion and 48 jours after.
To assess the minor complications of wearing the ARFC mask . | Hour: 48
  Occurrence of minor complications related to the wearing of the mask as reported for non-invasive ventilation (dry mouth, nose, conjunctivitis, skin lesions at the support point, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc PERROT, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No